CLINICAL TRIAL: NCT02885909
Title: The Effects of Glucose Control and Monitor on Inflammation in the Hospitalized Patients With Hyperglycemia
Brief Title: Inpatient Blood Glucose Control in Taichung Veterans General Hospital
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF16199B
Record Dates: First submitted 2016-08-26; First posted 2016-09-01 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: HYPERGLYCEMIA
Keywords: type 2 diabetes; inpatient; glucose control; continue glucose monitor
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulin protocal with CGM (Active Comparator): Insulin protocal with continue glucose monitor
  Interventions: Device: CONTINUE GLUCOSE MONITOR; Procedure: Insulin protocal
- Insulin protocal (Active Comparator): Insulin protocal with convential glucose monitor
  Interventions: Procedure: Insulin protocal
- Convential treatment (No Intervention): Convential insulin treatment and glucose monitor

INTERVENTIONS:
Device: CONTINUE GLUCOSE MONITOR — Continue glucose monitor
  Arms: Insulin protocal with CGM
Procedure: Insulin protocal — Using insulin protocal based on glucose monitor
  Arms: Insulin protocal; Insulin protocal with CGM

SUMMARY:
This study will be conducted in the ward of Taichung Veterans General Hospital. The patient with hyperglycemia in hospitalization will be enrolled by glucose management team.

DETAILED DESCRIPTION:
This study will be conducted in the ward of Taichung Veterans General Hospital. The type 2 diabetic patient with hyperglycemia in hospitalization are candidates. The glucose will be controlled using the insulin protocal based on the glucose monitor systems. We will assess the effects of insulin protocal and glucose monitor system on the inpatient with hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic inpatient
* Fasting glucose >140 mg/dl or random glucose >180 mg/dl

Exclusion Criteria:

* incooperative for glucose monitor
* refusal of insulin
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-09; Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Glucose target | 6 days
  The ratio of glucose less than 180 mg/dl

SECONDARY OUTCOMES:
Fasting glucose target | 6 days
  the ratio of fasting glucose less than 140 mg/dl
Hypoglycemia | times
  symptoms or less than 70
Vascular Cell Adhesion Molecule 1 (VCAM-1) | 6 days
  Inflammation
Brain-Derived Neurotrophic Factor (BDNF) | 6 days
  Psychological assessment
Orexin-A | 6 days
  Psychological assessment

CONTACTS AND LOCATIONS:
Overall Officials: I-Te Lee, MD,PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available